CLINICAL TRIAL: NCT02966860
Title: A Single-Dose Study Evaluating the Oral Pharmacokinetics of an Oxycodone/Acetaminophen Solution in Healthy Subjects Under Fasted Conditions
Brief Title: Single-Dose PK Study of an Oxycodone/Acetaminophen Solution in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MNK15141038
Record Dates: First submitted 2016-11-06; First posted 2016-11-17 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxycodone and acetaminophen (OC/APAP) (Experimental): Single 15 mL dose of oral solution of OC/APAP (total dose 15 mg oxycodone/975 mg acetaminophen)
  Interventions: Drug: Oral solution OC/APAP

INTERVENTIONS:
Drug: Oral solution OC/APAP

SUMMARY:
A single-dose study evaluating the oral PK of an oxycodone/apap solution in healthy subjects under fasted conditions

DETAILED DESCRIPTION:
An open-label, single-dose, single-center study evaluating the oral PK of an oxycodone/apap solutions in healthy subjects under fasted conditions

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adequately informed and understands the nature and risks of the study and must be able to provide a signature and date on the informed consent form (ICF).
* Subjects must have a health status of "healthy" assessed by the investigator, defined as no clinically significant deviation from normal in medical history, physical examination, and clinical laboratory determinations.
* Subjects must be males or nonpregnant, nonlactating females, between 18 and 55 years of age (inclusive) at time of the Screening Visit.
* Subjects must have a body mass index (BMI) ≥ 19.0 and ≤ 30.0 kg/m² with a minimum weight of 110 pounds for females and 130 pounds for males at the Screening Visit. The BMI will be calculated using the standard formula of weight (kg)/(height [m])2.
* Female subjects must have a negative serum pregnancy test at the Screening Visit and check-in to the study site. All female subjects who are biologically capable of having children must agree and commit to the use of 2 acceptable methods of birth control, defined as nonhormonal forms of contraception, condoms or diaphragms with spermicidal foam 14 days prior to check-in to the study site and for the duration of study participation. Unacceptable methods of birth control include abstinence, hormone-containing intrauterine devices, uterine ablation, hormonal forms of contraception, rhythm, and withdrawal methods. Female subjects who are not biologically capable of having children are defined as postmenopausal female subjects who have been amenorrheic for at least 12 consecutive months prior to the Screening Visit or are surgically sterile.
* Male subjects with reproductive potential must agree to use an acceptable method of contraception for the duration of the study (surgical sterilization [vasectomy] or condom with spermicide).
* Subjects must be able to communicate effectively with study personnel.
* Subjects must be able and willing to follow all protocol requirements and study restrictions.

Exclusion Criteria:

* A subjects is ineligible for the study if he or she meets any of the following criteria at the Screening Visit or at check-in to the study site:
* Subject is from a vulnerable population, as defined by the Code of Federal Regulations Title 45, Part 46, Section 46.111(b), including but not limited to employees (temporary, part-time, full time, etc.) or a family member of the research staff conducting the study, or of the sponsor, or of the clinical research organization, or of the institutional review board (IRB).
* Subject has a history of any drug allergy, hypersensitivity, or intolerance to any opioids, APAP, or naltrexone which, in the opinion of the investigator, would place the subject at particular risk and compromise the safety of the subject in the study.
* Subject has a positive test result for human immunodeficiency virus (HIV), hepatitis B (surface antigen), or hepatitis C virus antibody.
* Subject has a thyroid-stimulating hormone (TSH) value that is outside the reference range at the Screening Visit.
* Subject has donated or had significant loss of whole blood (480 mL or more) within 30 days, or plasma within 14 days, prior to the Screening Visit or plans to donate blood or plasma while enrolled in this study.
* Subject has smoked or used nicotine-containing products 6 months prior to the Screening Visit.
* Subject has current or recent (within 2 years of the Screening Visit) drug or alcohol abuse, as defined in Diagnostic and Statistical Manual of Mental Disorders Fifth Edition, Diagnostic Criteria for Drug and Alcohol Abuse.
* Subject has current or recent (within 3 months of the Screening Visit) gastrointestinal (GI) disease (including, but not limited to, peptic ulcer, diverticulitis, bowel obstructions, adhesions, malabsorption, paralytic ileus, gastritis, or diarrhea) or any GI surgery that could impact the absorption of study drug (including, but not limited to, cholecystectomy and gastric bypass or gastric band surgery).
* Subject had any major surgery within 3 months prior to the Screening Visit.
* Subject has a history, or laboratory evidence of, a bleeding or clotting disorder or condition.
* Subject is unable to tolerate venipuncture and/or venous access.
* Subject has any medical, psychiatric and/or social reason for exclusion, as determined by the investigator.
* Subject has a positive test result for drugs of abuse (minimum: opioids, barbiturates, cannabinoids, benzodiazepines, cocaine, amphetamine), cotinine, or alcohol at the Screening Visit or at check-in to the study site.
* Subject used any other investigational medicinal product (study drug) within 30 days prior to the Screening Visit and throughout the duration of the study or plans to participate in another clinical study while concurrently enrolled in this study.
* Subject has taken prescription drugs or over-the-counter (OTC) medications, vitamins, minerals, or dietary/herbal supplements (including grapefruit juice and grapefruit-containing products, St. John's wort and St. John's wort-containing products) within 14 days prior to check-in to the study site and throughout the duration of the study.
* Subject has a history of conditions which might be specifically contraindicated or require caution to be used during the administration of any drug in the study.
* Subject presents with a history of acute illness within 14 days prior to check-in to the study site and throughout the duration of the study.
* Subject has an electrocardiogram (ECG) parameter (confirmed by repeat evaluation) outside the following limits: PR ≥ 210 ms, QRS ≥ 120 ms, QT ≥ 500 ms; QT interval corrected for heart rate incorporating Bazett's formula (QTcB) ≥ 450 ms.
* Subject has other clinically significant ECG abnormalities, as assessed by the investigator.
* Subject has an oxygen saturation of < 95%.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve from time 0 to the time of the last quantifiable sample (AUC0-t) | 24 hours
Observed maximum plasma concentration | 24 hours
Observed time to maximum plasma concentration | 24 hours
Apparent elimination half-life | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States